CLINICAL TRIAL: NCT01949818
Title: A Randomized, Controlled Mutiple-center Clinical Research on the Treatment With Yangzhengxiaoji Capsule Combination Chemotherapy for III/IV Diffuse Large B Cell Lymphoma
Brief Title: Treatment of Diffuse Large B Cell Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, The director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx2011-4
Record Dates: First submitted 2013-09-20; First posted 2013-09-25 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — VAP-cyclo protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yangzhengxiaoji Capsule combined with CHOP regimen (Experimental): Yangzhengxiaoji Capsule combined with CHOP(Cyclophosphamide,Vincristine,Doxorubicin,Prednisone) regimen
  Interventions: Drug: Yangzhengxiaoji capsule combined with CHOP regimen
- CHOP regimen (Experimental): CHOP(Cyclophosphamide,Vincristine,Doxorubicin,Prednisone) regimen
  Interventions: Drug: CHOP regimen

INTERVENTIONS:
Drug: Yangzhengxiaoji capsule combined with CHOP regimen — Yangzhengxiaoji capsule combined with CHOP regimen(Yangzhengxiaoji capsule,Cyclophosphamide,Vincristine,Doxorubicin,Prednisone)Yangzhengxiaoji capsule ,1.56g,Tid,p.o,d7-21, Cyclophosphamide 750mg/d,ivgtt, d1;Vincristine,1.4g/m2,ivgtt, d1;Doxorubicin,50mg/m2,ivgtt,d1;Prednisone 60mg/m2,p.o, d1-5.
  Arms: Yangzhengxiaoji Capsule combined with CHOP regimen
Drug: CHOP regimen — CHOP regimen(Cyclophosphamide,Vincristine,Doxorubicin,Prednisone) Cyclophosphamide 750mg/d,ivgtt, d1;Vincristine,1.4g/m2,ivgtt, d1;Doxorubicin,50mg/m2,ivgtt,d1;Prednisone 60mg/m2,p.o, d1-5
  Arms: CHOP regimen

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Yangzhengxiaoji Capsule Combination Chemotherapy for III/IV Diffuse Large B Cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

- Age range 14-70 years old; ECOG performance status 0-2; Estimated survival time > 3 months Histological confirmed Diffuse large B cell lymphoma(III/IV) None of chemotherapy or radiotherapy has been previously used None of chemotherapy contraindication: hemoglobin ≥ 90 g/dl, neutrophil ≥ 1.5×109/L, platelet ≥ 100×109/L, ALT and AST ≤ 2×ULN, serum bilirubin ≤ 1.5×ULN, serum creatine ≤ 1.5×upper limitation of normal (ULN), Serum Albumin ≥ 30g/L At least one measurable lesion None of other serious diseases, cardiopulmonary function is normal Pregnancy test of women at reproductive age must be negative Patients could be followed up None of other relative treatments including the traditional Chinese medicine, immunotherapy,biotherapy except anti-bone metastasis therapy and other symptomatic treatments.

Exclusion Criteria:

* Disagreement on blood sample collection Patients allergic of any of drug in this regimen or with metabolic disorder Pregnant or lactating women Serious medical illness likely to interfere with participation Serious infection Primitive or secondary tumors of central nervous system Chemotherapy or radiotherapy contraindication The evidence of CNS metastasis History of peripheral nervous disorder or dysphrenia patients participating in other clinical trials patients taking other antitumor drugs patients estimated to be unsuitable by investigation

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to end of follow-up-phase (approximately 24 months)

SECONDARY OUTCOMES:
overall survival | up to the date of death (approximately 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi Zhang, Dr, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China